CLINICAL TRIAL: NCT02607046
Title: Post-revascularization Rehabilitation to Improve Function in Veterans With PAD
Brief Title: Exercise Rehabilitation in Veterans With PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F1927-P; I21RX001927 (NIH)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: rehabilitation; exercise training
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Exercise Training
  Interventions: Other: Exercise training
- NMES (Experimental): Neuromuscular Electrical Stimulation
  Interventions: Other: NMES

INTERVENTIONS:
Other: Exercise training — The exercise program includes supervised and home-based walking and strength exercise.
  Arms: Exercise
Other: NMES — This intervention consists of using neuromuscular electrical stimulation (NMES) as a form of passive exercise for muscles in the legs.
  Arms: NMES

SUMMARY:
Peripheral artery disease (PAD) results in blockages of arteries (blood vessels) and decreased blood flow to the legs. This may cause difficulty or pain with walking or other activities that use leg muscles. Exercise may help improve blood flow in the legs and improve the ability to walk. This research project will be conducted patients with PAD that require revascularization. The goal is to examine the effects of 3 months of exercise rehabilitation or neuromuscular stimulation on leg blood flow, physical function, quality of life and general health.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) and its associated declines in physical function impair quality of life (QOL) in nearly 20% of older Veterans and result in substantial VA health care costs. Revascularization addresses the anatomical pathology, but does not restore mobility function and QOL. Optimal therapy may require post-revascularization rehabilitation to address lingering defects in skeletal muscle that limit function; however, the current standard of care after revascularization does not include rehabilitation. Exercise training and neuromuscular electrical stimulation (NMES) may enhance function by increasing muscle perfusion to improve outcomes in older Veterans with PAD after revascularization.

The investigators will enroll Veterans (50-80 years of age) with PAD who are planned for percutaneous revascularization. Participants will complete research testing consisting of: a) Assessment of mobility function and QOL; and b) Treadmill tests to assess ambulatory capacity, and calf muscle perfusion. Participants will undergo screening prior to revascularization and will have baseline testing 2-3 weeks after revascularization. After post-revascularization testing, patients will be randomized to Exercise-only or NMES-only. After completion of the 3-month intervention, participants will repeat all tests to determine the effects of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral arterial disease; or ankle-brachial index <0.9.
* Planned to undergo endovascular revascularization within 6 months.

Exclusion Criteria:

* Cancer under active treatment
* Planned for lower extremity bypass surgery
* Body mass index > 45 kg/m2
* Critical limb ischemia or lower extremity gangrene

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Prior, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kundi R, Prior SJ, Addison O, Lu M, Ryan AS, Lal BK. Contrast-Enhanced Ultrasound Reveals Exercise-Induced Perfusion Deficits in Claudicants. J Vasc Endovasc Surg. 2017;2(1):9. doi: 10.21767/2573-4482.100041. Epub 2017 Mar 6. PMID 28691118
- [Result] Addison O, Prior SJ, Kundi R, Serra MC, Katzel LI, Gardner AW, Ryan AS. Sarcopenia in Peripheral Arterial Disease: Prevalence and Effect on Functional Status. Arch Phys Med Rehabil. 2018 Apr;99(4):623-628. doi: 10.1016/j.apmr.2017.10.017. Epub 2017 Nov 11. PMID 29138051
- [Result] Addison O, Kundi R, Ryan AS, Goldberg AP, Patel R, Lal BK, Prior SJ. Clinical relevance of the modified physical performance test versus the short physical performance battery for detecting mobility impairments in older men with peripheral arterial disease. Disabil Rehabil. 2018 Dec;40(25):3081-3085. doi: 10.1080/09638288.2017.1367966. Epub 2017 Aug 23. PMID 28835180
- [Result] Prior SJ, Chrencik MT, Christensen E, Kundi R, Ryan AS, Addison O, Lal BK. An exercise stress test for contrast-enhanced duplex ultrasound assessment of lower limb muscle perfusion in patients with peripheral arterial disease. J Vasc Surg. 2024 Feb;79(2):397-404. doi: 10.1016/j.jvs.2023.10.005. Epub 2023 Oct 14. PMID 37844848

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants enrolled; only 35 participants completed baseline testing and were randomized.
Groups:
- Exercise: Exercise Training
  Exercise training: The exercise program includes supervised treadmill walking and home-based walking exercise.
Period: Overall Study
Arm/Group | Exercise | NMES
Started | 22 | 13
Completed | 14 | 10
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | NMES | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (5.3) | 69.7 (7.5) | 67.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 21 | 12 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 12 | 34
Modified Physical Performance Test [Mean (Standard Deviation); unit: scores on a scale] — Test of Mobility Function (minimum score = 0; maximum score = 36; higher score associated with better outcome)
  scores on a scale | 30.8 (3.5) | 30.7 (3.0) | 30.8 (3.2)
Six-minute Walk Distance [Mean (Standard Deviation); unit: feet] — Test of Ambulatory Capacity
  feet | 1237 (328) | 1070 (325) | 1164 (330)
Muscle Perfusion Measured by Ultrasound Scan [Mean (Standard Deviation); unit: units on a scale] — Calf Muscle Perfusion assessed as digital video intensity from recorded ultrasound scans. Units are scale data with a minimum = 0 and no predetermined maximum. Higher score = more perfusion.
  units on a scale | 4.57 (1.98) | 3.90 (2.01) | 4.28 (1.90)

OUTCOME MEASURES:

1. Primary Outcome: Modified Physical Performance Test
Description: Test of Mobility Function (minimum score = 0; maximum score = 36; higher score associated with better outcome)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Exercise | NMES
Number analyzed (Participants) | 14 | 10
scores on a scale | 31.8 (5.2) | 32.3 (3.0)

2. Primary Outcome: Six-minute Walk Distance
Description: Test of ambulatory capacity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Exercise | NMES
Number analyzed (Participants) | 14 | 10
feet | 1295 (287) | 1193 (191)

3. Secondary Outcome: Muscle Perfusion Measured by Ultrasound Scan
Description: Calf Muscle Perfusion assessed as digital video intensity from recorded ultrasound scans. Units are scale data with a minimum = 0 and no predetermined maximum. Higher score = more perfusion.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | NMES
Number analyzed (Participants) | 14 | 10
units on a scale | 6.13 (4.75) | 4.59 (2.49)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Exercise | NMES
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/13
Other Adverse Events (participants affected / at risk) | 4/22 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=22) | NMES (N=13)
Chest Pain (Cardiac disorders) | 1 (1) | NA — Exertional chest pain. Brief hospitalization; no intervention required
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=22) | NMES (N=13)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Elevated Blood Glucose (Endocrine disorders) | 1 (1) | 0 (0)
Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Toe injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Toe wound unrelated to study
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Single bout of hypotension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02607046/Prot_SAP_000.pdf